CLINICAL TRIAL: NCT03971071
Title: A Phase 4, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Erenumab in Adults With Chronic Migraine and Medication Overuse Headache
Brief Title: A Study to Evaluate the Efficacy and Safety of Erenumab in Adults With Medication Overuse Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20170703; 2018-003342-16 (EudraCT Number)
Record Dates: First submitted 2019-05-23; First posted 2019-06-03 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Migraine Headache
Keywords: Chronic Migraine; Medication Overuse Headache
MeSH Terms: conditions — Migraine Disorders; Headache Disorders, Secondary | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): After participants complete the baseline period and are found eligible, they will be enrolled and randomized in a 1:1:1 ratio to either erenumab (70 mg or 140 mg) or placebo.
  Interventions: Drug: Placebo
- Erenumab 70 mg (Active Comparator): After participants complete the baseline period and are found eligible, they will be enrolled and randomized in a 1:1:1 ratio to either erenumab (70 mg or 140 mg) or placebo.
  Interventions: Drug: Erenumab 70 mg
- Erenumab 140 mg (Active Comparator): After participants complete the baseline period and are found eligible, they will be enrolled and randomized in a 1:1:1 ratio to either erenumab (70 mg or 140 mg) or placebo.
  Interventions: Drug: Erenumab 140 mg

INTERVENTIONS:
Drug: Erenumab 70 mg — Erenumab once every 4 weeks. Subcutaneous injection.
  Other Names: Aimovig
  Arms: Erenumab 70 mg
Drug: Erenumab 140 mg — Erenumab once every 4 weeks. Subcutaneous injection.
  Other Names: Aimovig
  Arms: Erenumab 140 mg
Drug: Placebo — Placebo once every 4 weeks. Subcutaneous injection.
  Arms: Placebo

SUMMARY:
Study 20170703 is a phase 4, randomized, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy and safety of erenumab against placebo in participants with chronic migraine (CM) who have a history of at least 1 preventive treatment failure and are diagnosed with medication overuse headache (MOH).

DETAILED DESCRIPTION:
Study 20170703 is a phase 4, randomized, double-blind, double-dummy, parallel-group, placebo-controlled study to evaluate the safety and efficacy of erenumab against placebo in a CM population with MOH and prior history of treatment failure. Participants will be enrolled based on fulfilment of the International Classification of Headache Disorders, 3rd Edition (ICHD-3) CM and MOH criteria and will not be advised to early discontinue acute medication.

Participants who successfully complete the 24-week double-blind treatment period (DBTP) of the study will be offered an opportunity to continue in an open-label treatment period (OLTP) of 28-weeks duration. Participants who received erenumab treatment during the DBTP will continue to receive the same erenumab dose during the OLTP. Participants who received placebo during the DBTP will be allocated in a 1:1 ratio to receive either erenumab 70 mg or 140 mg SC QM during the OLTP. All participants will remain blinded to their original DBTP treatment assignment.

ELIGIBILITY:
Eligibility criteria will be evaluated during the up to 3-week screening period (part 1) and a 4-week baseline period (part 2). At the end of baseline period, participants who successfully met eligibility criteria will be randomized on study.

Key Inclusion Criteria Part 1: To be assessed during the 3-week screening period, prior to the baseline period. Participants are eligible to be included in the study only if all of the following criteria apply:

* Participant has provided informed consent prior to initiation of any study-specific activities/procedures
* Age ≥ 18 years on entry into the study
* Documented history of migraine without aura and/or migraine with aura according to the ICHD-3 classification for ≥ 12 months at screening
* Documented history of CM for a minimal duration of 6 months before screening
* Current diagnosis of MOH
* History of treatment failure with at least 1 preventive treatment as defined as treatment discontinuation due to lack of efficacy, adverse event or general poor tolerability

Key Exclusion Criteria Part 1

Participants are excluded from the study if any of the following criteria apply:

Disease Related

* Age > 50 years at migraine onset or > 65 years at CM onset
* History of hemiplegic migraine, cluster headache or other trigeminal autonomic cephalalgia
* Current concomitant diagnosis of a secondary type of headache other than MOH
* No therapeutic response in prevention of migraine after an adequate therapeutic trial of > 3 preventive treatment categories
* Changes in drug regimen (ie, changes in dose or frequency of use) of an allowed migraine preventive medication within 2 months prior to start of baseline
* Received botulinum toxin in the head and/or neck region within 4 months prior to screening
* Documented history of treatment with an anti-calcitonin gene-related peptide product preventive treatment
* Anticipated to require any excluded medication/device or procedure during the study

Other Medical Conditions

* History or evidence of unstable or clinically significant medical condition that, in the opinion of the investigator or Amgen's physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion
* Evidence of "recreational use" of illicit drugs within 12 months prior to screening, based on medical records, self-report, or a positive drug test performed during screening.

Key Inclusion Criteria Part 2. To be assessed at the end of the baseline period and prior to enrollment into DBTP. Based on information collected through the electronic diary (eDiary) during the baseline period, the following requirements must be met:

-≥ 14 headache days during the 28-day baseline period out of which ≥ 8 headache days meet criteria as migraine days

* Observation of acute migraine medication overuse during the baseline period. Medication overuse at baseline is defined as:
* ≥ 10 days of combination treatment OR
* ≥ 10 days of short-acting opioids/opioid-containing medication OR
* ≥ 10 days of triptans, ergots, OR
* ≥ 15 days of nonsteroidal anti-inflammatory drugs or simple analgesics intake
* At least 2 acute headache medication days per week for each week with at least 5 diary days
* Demonstrated at least 80% compliance with the eDiary (eg, must complete eDiary items on at least 23 out of 28 days during the baseline period)

Key Exclusion Criteria Part 2

Study Procedures

* Changed or planning to change the dose of an allowed concomitant medication that may have migraine preventive effect during baseline period or post-randomization
* Unstable or clinically significant medical condition that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion

Contraception, pregnancy or breastfeeding

* Unwillingness to maintain acceptable contraception method, when applicable
* Evidence of pregnancy or breastfeeding per participant self-report, medical records or positivity on baseline pregnancy screening tests, through end of study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (94):
- United States (32):
  - Core Healthcare Group, Cerritos, California
  - Axiom Research, Colton, California
  - Clinical Research Institute, Los Angeles, California
  - The George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - Floridian Clinical Research LLC, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Saint Lukes Clinic, Meridian, Idaho
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - College Park Family Care Center, Overland Park, Kansas
  - Collective Medical Research, Prairie Village, Kansas
  - University of Kentucky, Lexington, Kentucky
  - DelRicht Research, New Orleans, Louisiana
  - Neurology Center of New England PC, Foxborough, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute Inc, Minneapolis, Minnesota
  - Citizens Memorial Healthcare, Bolivar, Missouri
  - Mercy Research, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dent Neurosciences Research Center, Amherst, New York
  - Onsite Clinical Solutions LLC, Charlotte, North Carolina
  - Clinical Trial Investigator Clinical Research Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Allegheny Health Network Cancer Institute at Mellon Pavilion, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc, Pittsburgh, Pennsylvania
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Texas Neurology, PA, Dallas, Texas
  - Wasatch Clinical Research LLC, Salt Lake City, Utah
  - Marshall University, Huntington, West Virginia
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
- Australia (2):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- Austria (4):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Konventhospital der Barmherzigen Brueder Linz, Linz
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Czechia (7):
  - Neurologie Brno sro, Brno
  - Fakultni nemocnice u svate Anny v Brne, Brno
  - Dado Medical sro, Prague
  - Thomayerova nemocnice, Prague
  - INEP, Prague
  - Mudr Stanislav Bartek sro, Přerov
  - Vestra Clinics sro, Rychnov nad Kněžnou
- Finland (4):
  - Helsingin Paansarkykeskus Aava, Helsinki
  - Northern Cinical Trial Coordinators, Oulu
  - Suomen Terveystalo, Tampere
  - Terveystalo Pulssi, Turku
- France (9):
  - Hospices Civils de Lyon - Hopital neurologique Pierre Wertheimer, Bron
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Roger Salengro, Lille
  - Hopital La Timone, Marseille
  - Centre Hospitalier Universitaire de Nice - Hopital de Cimiez, Nice
  - Hopital Lariboisiere, Paris
  - Groupe hospitalier Paris Saint Joseph, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Annecy Genevois, Pringy
  - Centre Hospitalier Universitaire Saint-Etienne - Hopital Nord, Saint-Etienne
- Hungary (7):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Swiss Premium Egeszsegkozpont, Budapest
  - Orszagos Mentalis, Ideggyogyaszati es Idegsebeszeti Intezet, Budapest
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz, Debrecen
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
- Italy (7):
  - IRCCS Istituto delle Scienze Neurologiche di Bologna Ospedale Bellaria, Bologna
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione Istituto Neurologico Nazionale C Mondino IRCCS, Pavia
  - IRCCS San Raffaele Pisana, Roma
- Poland (5):
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Spolka Jawna, Ksawerów
  - Jerzy Petz Mediq Niepubliczny Zaklad Opieki Zdrowotnej, Legionowo
  - Gabinet Lekarski Jacek Rozniecki, Lodz
  - Clinical Research Center Spzoo Medic-R Spolka Komandytowa, Poznan
  - RCMed Oddzial Sochaczew, Sochaczew
- Portugal (4):
  - Hospital Professor Doutor Fernando Fonseca, EPE, Amadora
  - Hospital da Luz, SA, Lisbon
  - Centro Hospitalar de Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
  - Campus Neurologico Senior, Torres Vedras
- Spain (7):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Clinico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
- United Kingdom (6):
  - Queen Elizabeth University Hospital, Glasgow
  - Hull Royal Infirmary, Hull
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Kings College London, London
  - Royal Victoria Infirmary, Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Tepper SJ, Dodick DW, Lanteri-Minet M, Dolezil D, Gil-Gouveia R, Lucas C, Piasecka-Stryczynska K, Szabo G, Mikol DD, Chehrenama M, Chou DE, Yang Y, Paiva da Silva Lima G. Efficacy and Safety of Erenumab for Nonopioid Medication Overuse Headache in Chronic Migraine: A Phase 4, Randomized, Placebo-Controlled Trial. JAMA Neurol. 2024 Sep 16;81(11):1140-9. doi: 10.1001/jamaneurol.2024.3043. Online ahead of print. PMID 39283627
- [Background] Tepper SJ, Dodick DW, Lanteri-Minet M, Dolezil D, Gil-Gouveia R, Lucas C, Piasecka-Stryczynska K, Szabo G, Mikol DD, Chehrenama M, Chou DE, Liu Z, da Silva Lima GP. Efficacy and Safety of Erenumab in Adults With Medication Overuse Headache: Final Results From a Phase 4 Randomized Placebo-Controlled Study. Eur J Neurol. 2025 Aug;32(8):e70328. doi: 10.1111/ene.70328. PMID 40838472
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 67 study centers in North America, Europe, and Australia, and participated from 07 October 2019 to 13 June 2023.
Pre-assignment Details: Adult participants with a history of chronic migraine and medication overuse headaches according to the International Classification of Headache Disorders 3rd Edition (ICHD-3) criteria were randomized 1:1:1 to receive erenumab 70 mg or 140 mg subcutaneously (SC) once every 4 weeks (QM) or matching placebo. Prior to randomization, participants completed a 4-week baseline period to evaluate eligibility.
Groups:
- Placebo (DBTP): Participants were randomized to receive matching placebo SC QM for 24 weeks in the DBTP.
- Erenumab 70 mg (DBTP): Participants were randomized to receive 1 mL of erenumab 70 mg/mL SC QM for 24 weeks in the DBTP.
- Erenumab 140 mg (DBTP): Participants were randomized to receive 1 mL of erenumab 140 mg/mL SC QM for 24 weeks in the DBTP.
- Erenumab 70 mg (OLTP): Eligible participants who successfully completed the DBTP continued to the Open-label Treatment Period (OLTP) and received erenumab 70 mg SC QM for up to 28 weeks (up to Week 52).
  Eligible participants included participants randomized to erenumab 70 mg in the DBTP and participants randomized to placebo in the DBTP, re-randomized to erenumab 70 mg in the OLTP.
- Erenumab 140 mg (OLTP): Eligible participants who successfully completed the DBTP continued to the OLTP and received erenumab 140 mg SC QM for up to 28 weeks (up to Week 52).
  Eligible participants included participants randomized to erenumab 140 mg in the DBTP and participants randomized to placebo in the DBTP, re-randomized to erenumab 140 mg in the OLTP.
Period: Double-blind Treatment Period (DBTP)
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP) | Erenumab 70 mg (OLTP) | Erenumab 140 mg (OLTP)
Started | 206 | 207 | 207 | 0 | 0
Opioid-treated Cohort (> 4 days/month opioid medication use in baseline period; included for purposes of exploratory analyses only) | 12 | 12 | 12 | 0 | 0
Nonopioid-treated Cohort (≤ 4 days/month opioid medication use in baseline period) | 194 | 195 | 195 | 0 | 0
Completed (Completed DBTP (Week 24)) | 197 | 193 | 201 | 0 | 0
Not Completed | 9 | 14 | 6 | 0 | 0
Not completed — Sponsor decision | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 11 | 6 | 0 | 0
Not completed — Other | 2 | 2 | 0 | 0 | 0
Period: Open-label Treatment Period
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP) | Erenumab 70 mg (OLTP) | Erenumab 140 mg (OLTP)
Started | 0 | 0 | 0 | 291 | 296
Completed | 0 | 0 | 0 | 281 | 281
Not Completed | 0 | 0 | 0 | 10 | 15
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 10 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP) | Total
Number analyzed (Participants) | 206 | 207 | 207 | 620
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (12.5) | 43.1 (11.6) | 43.5 (12.2) | 43.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 170 | 174 | 510
  Male | 40 | 37 | 33 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 13 | 32
  Not Hispanic or Latino | 196 | 197 | 194 | 587
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 2 | 8
  White | 196 | 187 | 187 | 570
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 15 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of Medication Overuse Headaches (MOH) at Month 6
Description: Absence of MOH at month 6 was defined as mean monthly acute headache medication days (AHMD) < 10 days over months 4, 5, and 6 (weeks 13 through 24) or mean monthly headache days < 14 days over months 4, 5, and 6 (weeks 13 through 24) of the DBTP where an AHMD was defined as a calendar day in which the participant took at least 1 acute headache medication.
Time Frame: Months 4, 5, and 6 (weeks 13 through 24) of the DBTP
Population: Efficacy analysis set (nonopioid-treated cohort): randomized participants with an opioid medication use of ≤ 4 days per month during the baseline period and who received at least 1 dose of IP during DBTP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP)
Number analyzed (Participants) | 194 | 194 | 194
Participants | 102 | 117 | 134
Statistical Analysis 1: Comparison: Placebo (DBTP) vs Erenumab 70 mg (DBTP); Test type: Superiority; p = 0.13, Cochran-Mantel-Haenszel; Common odds ratio = 1.37, 95% CI 2-sided [0.92 to 2.05] — Erenumab 70 mg versus Placebo. Common odds ratio and p-value were obtained from a Cochran-Mantel-Haenszel test, stratified by concomitant oral migraine preventive treatment initiated before screening and taken during baseline (Yes or No)
Statistical Analysis 2: Comparison: Placebo (DBTP) vs Erenumab 140 mg (DBTP); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Common odds ratio = 2.01, 95% CI 2-sided [1.33 to 3.05] — Erenumab 140 mg versus Placebo. Common odds ratio and p-value were obtained from a Cochran-Mantel-Haenszel test, stratified by concomitant oral migraine preventive treatment initiated before screening and taken during baseline (Yes or No)

2. Secondary Outcome: Change From Baseline in Mean Monthly AHMDs Over Months 4, 5, and 6
Description: An AHMD was defined as a calendar day in which the participant takes at least 1 acute headache medication. Acute headache medications included triptan-based, ergotamine-based and ditan-based migraine medications, non-opioid and opioid-containing acute headache medications, non-opioid butalbital and opioid-containing butalbital containing medications.
Time Frame: Baseline and months 4, 5, and 6 (weeks 13 through 24) of the DBTP
Population: Efficacy analysis set (nonopioid-treated cohort): randomized participants with an opioid medication use of ≤ 4 days per month during the baseline period and who received at least 1 dose of IP during DBTP. Participants with evaluable data from weeks 13 through 24 are included.
Measure: Least Squares Mean (Standard Error); unit: days per month
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP)
Number analyzed (Participants) | 194 | 193 | 194
days per month | -6.61 (0.41) | -7.83 (0.41) | -9.35 (0.41)
Statistical Analysis 1: Comparison: Placebo (DBTP) vs Erenumab 70 mg (DBTP); Test type: Superiority; p = 0.033, Linear Mixed Model — Nominal p-value is presented without multiplicity adjustment; Least squares mean difference = -1.23, 95% CI 2-sided [-2.35 to -0.10] — Erenumab 70 mg versus Placebo. Covariates: treatment, visit, treatment-by-visit, concomitant oral migraine preventive treatment initiated before screening and taken during baseline (Yes or No), and baseline value
Statistical Analysis 2: Comparison: Placebo (DBTP) vs Erenumab 140 mg (DBTP); Test type: Superiority; p < 0.001, Linear Mixed Model — Nominal p-value is presented without multiplicity adjustment; Least squares mean difference = -2.74, 95% CI 2-sided [-3.87 to -1.62] — Erenumab 140 mg versus Placebo. Covariates: treatment, visit, treatment-by-visit, concomitant oral migraine preventive treatment initiated before screening and taken during baseline (Yes or No), and baseline value

3. Secondary Outcome: Number of Participants With Sustained MOH Remission at Month 6
Description: Sustained MOH remission was defined as the absence of MOH at month 3 (week 12) and month 6 (week 24) of the DBTP. Absence of MOH was achieved when mean monthly AHMD < 10 days or mean monthly headache days < 14 days over the 3-month period (weeks 12 to 24).
Time Frame: Month 3 (week 12) to month 6 (week 24) of the DBTP
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP)
Number analyzed (Participants) | 194 | 194 | 194
Participants | 73 | 96 | 119
Statistical Analysis 1: Comparison: Placebo (DBTP) vs Erenumab 70 mg (DBTP); Test type: Superiority; p = 0.019, Cochran-Mantel-Haenszel; Common odds ratio = 1.62, 95% CI 2-sided [1.08 to 2.43] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo (DBTP) vs Erenumab 140 mg (DBTP); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Common odds ratio = 2.63, 95% CI 2-sided [1.75 to 3.96] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Change From Baseline in Mean Monthly Average Physical Impairment Domain Scores as Measured by the Migraine Physical Function Impact Diary (MPFID)
Description: The MPFID is a self-administered 13-item instrument measuring physical functioning, completed daily using the eDiary. The physical impairment domain includes 5 items. Participants respond to items using a 5-point scale, with difficulty items ranging from "Without any difficulty" to "Unable to do", and frequency items ranging from "None of the time" to "All of the time". Each item is assigned a score from 1 to 5, with 5 representing the greatest burden. For each domain, the scores are calculated as the sum of the item responses and the sum is rescaled to a 0 to 100 scale, with higher scores representing greater impact of migraine, i.e., higher burden.
Time Frame: Baseline and months 4, 5, and 6 (weeks 13 through 24) of the DBTP
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP)
Number analyzed (Participants) | 194 | 193 | 194
Scores on a scale | -8.50 (0.86) | -11.75 (0.87) | -10.63 (0.86)
Statistical Analysis 1: Comparison: Placebo (DBTP) vs Erenumab 70 mg (DBTP); Test type: Superiority; p = 0.007, Linear Mixed Model — Nominal p-value is presented without multiplicity adjustment; Least squares mean difference = -3.25, 95% CI 2-sided [-5.62 to -0.88] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo (DBTP) vs Erenumab 140 mg (DBTP); Test type: Superiority; p = 0.075, Linear Mixed Model — Nominal p-value is presented without multiplicity adjustment; Least squares mean difference = -2.13, 95% CI 2-sided [-4.48 to 0.22] — [estimate comment as in outcome 2, analysis 2]

5. Secondary Outcome: Change From Baseline in Mean Monthly Average Impact on Everyday Activities Domain Scores as Measured by the MPFID
Description: The MPFID is a self-administered 13-item instrument measuring physical functioning, completed daily using the eDiary. The impact on everyday activities domain includes 7 items. Participants respond to items using a 5-point scale, with difficulty items ranging from "Without any difficulty" to "Unable to do", and frequency items ranging from "None of the time" to "All of the time". Each item is assigned a score from 1 to 5, with 5 representing the greatest burden. For each domain, the scores are calculated as the sum of the item responses and the sum is rescaled to a 0 to 100 scale, with higher scores representing greater impact of migraine, i.e., higher burden.
Time Frame: Baseline and months 4, 5, and 6 (weeks 13 through 24) of the DBTP
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP)
Number analyzed (Participants) | 194 | 193 | 194
Scores on a scale | -10.91 (0.84) | -13.52 (0.85) | -13.29 (0.84)
Statistical Analysis 1: Comparison: Placebo (DBTP) vs Erenumab 70 mg (DBTP); Test type: Superiority; p = 0.028, Linear Mixed Model — Nominal p-value is presented without multiplicity adjustment; Least squares mean difference = -2.61, 95% CI 2-sided [-4.92 to -0.29] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo (DBTP) vs Erenumab 140 mg (DBTP); Test type: Superiority; p = 0.043, Linear Mixed Model — Nominal p-value is presented without multiplicity adjustment; Least squares mean difference = -2.37, 95% CI 2-sided [-4.67 to -0.07] — [estimate comment as in outcome 2, analysis 2]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse event (AE) that started on or after first dose of IP, and up to the end of the study (52 weeks).
  Any clinically significant changes in vital signs were included as TEAEs.
Time Frame: Day 1 to Week 24 (DBTP) and Week 25 to 52 weeks (OLTP)
Population: Safety analysis set: randomized participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Groups:
- Erenumab 70 mg (OLTP): Eligible participants who successfully completed the DBTP continued to the OLTP and received erenumab 70 mg SC QM for up to 28 weeks (up to Week 52).
  Eligible participants included participants randomized to erenumab 70 mg in the DBTP and participants randomized to placebo in the DBTP, re-randomized to erenumab 70 mg in the OLTP.
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP) | Erenumab 70 mg (OLTP) | Erenumab 140 mg (OLTP)
Number analyzed (Participants) | 206 | 206 | 206 | 291 | 296
Participants | 130 | 139 | 142 | 178 | 182

ADVERSE EVENTS:
Time Frame: Day 1 to Week 24 (DBTP) and Week 25 to 52 weeks (OLTP).
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Placebo (DBTP) | Erenumab 70 mg (DBTP) | Erenumab 140 mg (DBTP) | Erenumab 70 mg (OLTP) | Erenumab 140 mg (OLTP)
All-Cause Mortality (participants affected / at risk) | 0/206 | 0/207 | 0/207 | 0/291 | 0/296
Serious Adverse Events (participants affected / at risk) | 8/206 | 3/206 | 3/206 | 6/291 | 12/296
Other Adverse Events (participants affected / at risk) | 29/206 | 67/206 | 72/206 | 65/291 | 75/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (DBTP) (N=206) | Erenumab 70 mg (DBTP) (N=206) | Erenumab 140 mg (DBTP) (N=206) | Erenumab 70 mg (OLTP) (N=291) | Erenumab 140 mg (OLTP) (N=296)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Embolic pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Intestinal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (DBTP) (N=206) | Erenumab 70 mg (DBTP) (N=206) | Erenumab 140 mg (DBTP) (N=206) | Erenumab 70 mg (OLTP) (N=291) | Erenumab 140 mg (OLTP) (N=296)
Constipation (Gastrointestinal disorders) | 9 | 31 | 34 | 22 | 24
COVID-19 (Infections and infestations) | 14 | 25 | 33 | 31 | 39
Nasopharyngitis (Infections and infestations) | 4 | 12 | 9 | 15 | 14
Insomnia (Psychiatric disorders) | 4 | 8 | 12 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03971071/Prot_002.pdf
  • Statistical Analysis Plan (2022-12-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03971071/SAP_003.pdf